CLINICAL TRIAL: NCT01642186
Title: A Randomized Three Arm Phase II Study of (1) Everolimus, (2) Estrogen Deprivation Therapy (EDT) With Leuprolide + Letrozole and (3) Everolimus + EDT in Patients With Unresectable Fibrolamellar Hepatocellular Carcinoma (FLL-HCC)
Brief Title: Study of (1) Everolimus, (2) Estrogen Deprivation Therapy (EDT) With Leuprolide + Letrozole and (3) Everolimus + EDT in Patients With Unresectable Fibrolamellar Hepatocellular Carcinoma (FLL-HCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Fibrolamellar Cancer Foundation (Other); Dana-Farber Cancer Institute (Other); Johns Hopkins University (Other); University of California, San Francisco (Other); Abbott (Industry); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 11-211
Record Dates: First submitted 2012-07-12; First posted 2012-07-17 (Estimated); Results first posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2021-07

CONDITIONS: Fibrolamellar Carcinoma; Fibrolamellar Liver Cancer
Keywords: LETROZOLE; LUPRON DEPOT; RAD001 (EVEROLIMUS); 11-211
MeSH Terms: conditions — Fibrolamellar hepatocellular carcinoma | interventions — Everolimus; Letrozole; Leuprolide

ARMS (3):
- Arm A everolimus (Experimental): Everolimus will be administered at the following doses:
  * Patients with a BSA ≤ 1.5 m2 will receive everolimus 5 mg PO QD.
  * Patients with a BSA > than or = to 1.5 m2 will receive everolimus 7.5 mg PO QD. If the patient is randomized to everolimus alone (1) or leuprolide and letrozole (2) and the cancer continues to grow, they may have the option to receive all three drugs together.
  Interventions: Drug: everolimus
- Arm B letrozole plus leuprolide (Experimental): Day 1 of Cycle 1: Leuprolide 7.5 mg IM will be administered by a nurse in clinic.
  Letrozole will be dispensed and will be taken at home. Patients will be instructed to take letrozole at the same time each day, consistently with food or without food, and swallowed whole with a glass of water. If the patient is randomized to everolimus alone (1) or leuprolide and letrozole (2) and the cancer continues to grow, they may have the option to receive all three drugs together.
  Interventions: Drug: letrozole plus leuprolide
- Arm C combination everolimus, letrozole and leuprolide (Experimental): * Patients with a BSA ≤ 1.5 m2 will receive everolimus 5 mg PO QD.
  * Patients with a BSA > than or = to 1.5 m2 will receive everolimus 7.5 mg PO QD. Leuprolide 7.5 mg IM will be given every 4 weeks (+/- 7 days). Everolimus and letrozole will be administered continuously using the same dose, schedule and administration. Everolimus, letrozole and leuprolide should be administered concurrently at all times.
  Interventions: Drug: combination of everolimus, letrozole and leuprolide

INTERVENTIONS:
Drug: everolimus
  Arms: Arm A everolimus
Drug: letrozole plus leuprolide
  Arms: Arm B letrozole plus leuprolide
Drug: combination of everolimus, letrozole and leuprolide
  Arms: Arm C combination everolimus, letrozole and leuprolide

SUMMARY:
There is no effective standard treatment for fibrolamellar liver cancer that cannot be removed by surgery. The investigators want to find out what effects, good and/or bad, 3 drugs called letrozole, leuprolide and everolimus will have on cancer. All of these drugs are FDA approved for the treatment of different cancers. Letrozole and leuprolide stop the body from producing estrogen, a normal hormone produced by the body. Too much estrogen may help fibrolamellar liver cancer grow. Everolimus is a drug that may block other chemicals in the body that can help cancer grow. The combination of letrozole and leuprolide plus everolimus may work well together.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 12 years old.
* Pathologically confirmed diagnosis of advanced and/or unresectable FLL-HCC. This will be performed by the participating centers on submitted specimens. If the submitted material is insufficient for analysis, a repeat biopsy is recommended.
* ECOG performance status 0-2 ; Lansky performance score of ≥ 60% for patients 12-16 years old
* Adequate hematologic, renal and hepatic function defined as:

Hematologic: ANC ≥ 1.0 x 10^9/L, platelets ≥ 50 x 10^9/L o Renal: creatinine ≤ 2 x upper limit of normal, or creatinine Clearance of ≥60 cc/mL/1.73 m^2 for patients > 16 years old. For patients ≤ 16 years of age, creatinine Clearance of ≥70 cc/mL/1.73 m^2 or serum creatinine based on the following chart: Creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73 m^2 or serum creatinine based on age/gender as follows: Age Maximum Serum Creatinine (mg/dL) Male Female 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4

≥ 16 years 1.7 1.4 The threshold creatinine values in this Table were derived from the Schwartz formula for estimating GFR (Schwartz et al. J. Peds, 106:522, 1985) utilizing child length and stature data published by the CDC.

* Hepatic: total bilirubin ≤ 2 mg/dL, alanine and aminotransferase levels ≤ 5 x upper limit of normal for age.
* Fasting blood glucose <1.5 x upper limit of normal . If fasting glucose > 1.5 x upper limit of normal, adequate glycemic control (fasting glucose < 1.5 x upper limit of normal ) for three weeks is recommended before starting protocol therapy.

  * At least 1 target lesion measurable by Response Evaluation Criteria in Solid Tumors (RECIST 1.1) guidelines.
* Target lesion(s) must not lie within a previously resected, irradiated, ablated, or chemoembolized area. If a lesion does lie in such an area, there must be evidence of a ≥ 20% increase in diameter and/or the appearance of a new lesion on subsequent imaging in order for such a lesion to be considered a target lesion.

  * Prior systemic therapy is allowed. Prior surgery, locoregional ablative or embolic therapies are also permitted provided that the criteria for measurable disease as outlined above are met.
  * Concurrent antiviral therapy for hepatitis B is permitted
  * Women of childbearing potential must be practicing an effective method of birth control that may include intrauterine devices (both hormonal and non-hormonal are acceptable), double-barrier method, male partner sterilization or abstinence, before enrollment, and throughout the study and for 6 months after receiving the last dose of study drug.
  * Men must agree to use a double barrier method of birth control and to not donate sperm during the study and for 6 months after receiving the last dose of study drugs. Sperm banking is acceptable for interested male patients enrolled on study prior to initiating treatment. Prescription oral contraceptives, contraceptive injections, and contraceptive patch are not approved methods of contraception in this study.
  * Negative pregnancy test (serum hCG) result (applicable to women of child bearing potential) within 7 days before Cycle 1 Day 1 of study treatment.

Exclusion Criteria:

* Concurrent anticancer, or radiation therapy. Patients must have completed all anticancer therapy > 4 weeks before the start of study therapy. The date of last palliative radiation must be > 2 weeks from the start of study therapy. Palliative radiation is permitted on protocol with MSK PI discretion on treatment modifications.
* Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) .
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* Concurrent oral contraceptive use or hormonal replacement therapy.
* Use of an aromatase inhibitor, GnRH agonist and/or tamoxifen within the past 30 days. Patients previously on fulvestrant or a q3 month GnRH agonist must have discontinued these medications for at least 3 months.
* Concurrent use of potent CYP3A4 and/or P-glycoprotein inhibitors or potent CYP3A4 inducers (please see Appendices 3 and 4). Where possible, otherwise eligible patients should be switched to alternative agents; otherwise, they will be excluded from the study.
* Potent CYP3A4 inducers decrease serum everolimus levels and should not be given concomitantly. Dose modifications of everolimus are not indicated in the presence of moderate CYP3A4 inducers [108]. Please refer to Appendix 3 for a complete list of potent and moderate inducers of CYP3A4.
* Potent CYP3A4 and/or P-glycoprotein inhibitors can increase serum levels of everolimus and should not be co-administered. Moderate inhibitors may mildly-moderately increase serum everolimus levels, though there is no definitive evidence supporting a dose reduction [108]. Please refer to Appendix 4 for a complete list of potent and moderate inhibitors of CYP3A4.
* Any investigational drug received within one month of study enrollment.
* Any severe, uncontrolled medical conditions that, in the opinion of the investigator, may be exacerbated by study therapy including infection, diabetes and cardiopulmonary disease.
* Any psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or nursing women.
* Patients with a known hypersensitivity to everolimus, letrozole, leuprolide and/or related compounds or their excipients.
* Patients who received any form of transplant and who are on any form of immunosuppressive therapy. However transplanted patients who are off immunosuppressive therapy for at least 4 weeks are allowed on the study, provided that any of their immunosuppressive-related toxicities have recovered to at least a grade 1.
* Known HIV positive with a CD4 count < 500 cells/mm3.
* Immunization with a live vaccine < 1 week of initiating study therapy or during therapy.
* BSA <1 m^2

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-07-12 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ghassan Abou-Alfa, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - University of California San Francisco, San Francisco, California
  - John Hopkins Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Derived] Lim II, Farber BA, LaQuaglia MP. Advances in fibrolamellar hepatocellular carcinoma: a review. Eur J Pediatr Surg. 2014 Dec;24(6):461-6. doi: 10.1055/s-0034-1396420. Epub 2014 Dec 8. PMID 25486412
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A Everolimus: Everolimus will be administered at the following doses:
  * Patients with a BSA ≤ 1.5 m2 will receive everolimus 5 mg PO QD.
  * Patients with a BSA > than or = to 1.5 m2 will receive everolimus 7.5 mg PO QD. If the patient is randomized to everolimus alone (1) or leuprolide and letrozole (2) and the cancer continues to grow, they may have the option to receive all three drugs together.
  everolimus
- Arm B Letrozole Plus Leuprolide: Day 1 of Cycle 1: Leuprolide 7.5 mg IM will be administered by a nurse in clinic.
  Letrozole will be dispensed and will be taken at home. Patients will be instructed to take letrozole at the same time each day, consistently with food or without food, and swallowed whole with a glass of water. If the patient is randomized to everolimus alone (1) or leuprolide and letrozole (2) and the cancer continues to grow, they may have the option to receive all three drugs together.
  letrozole plus leuprolide
- Arm C Combination Everolimus, Letrozole and Leuprolide: * Patients with a BSA ≤ 1.5 m2 will receive everolimus 5 mg PO QD.
  * Patients with a BSA > than or = to 1.5 m2 will receive everolimus 7.5 mg PO QD. Leuprolide 7.5 mg IM will be given every 4 weeks (+/- 7 days). Everolimus and letrozole will be administered continuously using the same dose, schedule and administration. Everolimus, letrozole and leuprolide should be administered concurrently at all times.
  combination of everolimus, letrozole and leuprolide
Period: Overall Study
Arm/Group | Arm A Everolimus | Arm B Letrozole Plus Leuprolide | Arm C Combination Everolimus, Letrozole and Leuprolide
Started | 9 | 9 | 10
Completed | 9 | 7 | 7
Not Completed | 0 | 2 | 3
Not completed — Death | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A Everolimus | Arm B Letrozole Plus Leuprolide | Arm C Combination Everolimus, Letrozole and Leuprolide | Total
Number analyzed (Participants) | 9 | 9 | 10 | 28
Age, Continuous [Mean (Full Range); unit: years] | 26 [21 to 50] | 27 [16 to 41] | 29 [20 to 45] | 27 [16 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 5 | 14
  Male | 5 | 4 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 9 | 10 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 8 | 8 | 8 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 9 | 10 | 28

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Endpoints for Part 1 of the Study is Progression-free Survival at 6 Months (PFS6)
Description: for Part 1 of the study is progression-free survival at 6 months (PFS6). A progression event refers to the first evidence of radiographic disease progression, clinical progression as determined by study investigators, or death. Imaging performed in 6 months will be used to determine PFS6.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A Everolimus | Arm B Letrozole Plus Leuprolide | Arm C Combination Everolimus, Letrozole and Leuprolide
Number analyzed (Participants) | 9 | 9 | 10
Participants
  Progression Free | 0 | 0 | 0
  Participants With Progression | 9 | 9 | 10

2. Secondary Outcome: Median PFS
Description: Kaplan-Meier PFS will be measured from the date that study therapy is initiated until the date of first evidence of radiographic disease progression, global clinical deterioration as determined by study investigators, or death.
Time Frame: 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Arm A Everolimus | Arm B Letrozole Plus Leuprolide | Arm C Combination Everolimus, Letrozole and Leuprolide
Number analyzed (Participants) | 9 | 9 | 10
months | 2.6 [0.9 to 5.5] | 2.7 [1.7 to 5.2] | 2.4 [1.0 to 2.9]

3. Secondary Outcome: Median Overall Survival (OS)
Description: Kaplan-Meier OS will be measured from the date that study therapy was commenced until the date of death.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
Measure: Median (Full Range); unit: months
Arm/Group | Arm A Everolimus | Arm B Letrozole Plus Leuprolide | Arm C Combination Everolimus, Letrozole and Leuprolide
Number analyzed (Participants) | 9 | 9 | 10
months | 12.5 [2.7 to 41.9] | 14.0 [3.2 to 22.4] | 10.6 [2.3 to 20.9]

4. Secondary Outcome: Percentage of Participants With Stable Disease
Description: Objective responses will be reported using RECIST guidelines (version 1.1). Objective response will be estimated using binomial proportions and exact 95% CIs will be provided. Stable Disease is defined as neither sufficient shrinkage (compared to baseline) to qualify for Partial Reponse nor sufficient increase (taking as reference the smallest sum diameters while on study) to qualify for Progressive Disease.
Time Frame: 2 years
Measure: Number; unit: Percentage of pts with stable disease
Arm/Group | Arm A Everolimus | Arm B Letrozole Plus Leuprolide | Arm C Combination Everolimus, Letrozole and Leuprolide
Number analyzed (Participants) | 9 | 9 | 10
Percentage of pts with stable disease | 55 | 37 | 11

5. Secondary Outcome: Number of Participants With One or More Adverse Events/Toxicity
Description: Adverse events/toxicity will be monitored and recorded using the CTCAE version 4.0 and summarized descriptively.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A Everolimus | Arm B Letrozole Plus Leuprolide | Arm C Combination Everolimus, Letrozole and Leuprolide
Number analyzed (Participants) | 9 | 9 | 10
Participants | 9 | 9 | 10

6. Secondary Outcome: Number of Participants With Tissue Biomarkers Collected
Description: Associations between baseline tissue biomarkers and PFS6 will be assessed using Fisher's exact test for categorical biomarkers, trend tests for ordinal biomarkers and Wilcoxon rank-sum test for continuous biomarkers. For patients undergoing surgery, changes in tissue biomarkers from baseline to surgery will be summarized descriptively in an exploratory fashion.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A Everolimus | Arm B Letrozole Plus Leuprolide | Arm C Combination Everolimus, Letrozole and Leuprolide
Number analyzed (Participants) | 9 | 9 | 10
Participants | 9 | 9 | 10

ADVERSE EVENTS:
Time Frame: Up to 100 months
Arm/Group | Arm A Everolimus | Arm B Letrozole Plus Leuprolide | Arm C Combination Everolimus, Letrozole and Leuprolide
All-Cause Mortality (participants affected / at risk) | 0/9 | 2/9 | 2/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 9/9 | 9/9 | 9/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A Everolimus (N=9) | Arm B Letrozole Plus Leuprolide (N=9) | Arm C Combination Everolimus, Letrozole and Leuprolide (N=10)
ALT increased (Investigations) | 7 | 7 | 8
Alkaline phosphatase increased (Investigations) | 7 | 8 | 9
Anemia (Blood and lymphatic system disorders) | 4 | 8 | 8
AST increased (Investigations) | 8 | 8 | 8
Blood bilirubin increased (Investigations) | 0 | 3 | 3
Cholesterol high (Investigations) | 5 | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Fatigue (General disorders) | 8 | 8 | 6
Mucositis oral (Gastrointestinal disorders) | 3 | 1 | 3
Nausea (Gastrointestinal disorders) | 3 | 4 | 5
Neutrophil count decreased (Investigations) | 0 | 1 | 3
Platelet count decreased (Investigations) | 3 | 2 | 6
Vomiting (Gastrointestinal disorders) | 3 | 5 | 4
White blood cell decreased (Investigations) | 3 | 3 | 7
Hypertriglyceridemia (Metabolism and nutrition disorders) | 6 | 3 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 5 | 8
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Death - NOS (General disorders) | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-12): https://cdn.clinicaltrials.gov/large-docs/86/NCT01642186/Prot_SAP_000.pdf